CLINICAL TRIAL: NCT07157371
Title: Effects of Supervised Structured Aerobic Exercise Training Program on Serum BDNF, Androgens Level, Menstrual Irregularity and Quality of Life in Females With Insulin Resistant Polycystic Ovarian Syndrome
Brief Title: Effects of Aerobic Exercise Training Program in Females With Insulin Resistant Polycystic Ovarian Syndrome
Acronym: SSAET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Muzna Munir, Assistant Professor, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC/RCR/ & AHS/23/1103
Record Dates: First submitted 2025-08-03; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovarian Syndrome (PCOS); Aerobic Exercise; Walking
Keywords: Insulin resistant; Supervised; aerobic exercise; SSAET; PCOS; metabolic syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome | interventions — Exercise; Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group- PCOS (Experimental): 25 weeks of supervised structured aerobic exercise treatment program will be applied on the females with PCOS in the gym setting.
  Interventions: Other: Supervised structured aerobic exercise training
- Second group- PCOS (Active Comparator): walk will be asked for these patients and their feedback will be taken through cell phone
  Interventions: Other: Walk

INTERVENTIONS:
Other: Supervised structured aerobic exercise training — Supervised structured aerobic exercise plan will be conducted in gym by the physiotherapist
  Other Names: Aerobic exercises
  Arms: Interventional group- PCOS
Other: Walk — Females with PCOS will be instructed to do a walk at home with medications
  Arms: Second group- PCOS

SUMMARY:
Design: RCT Randomized Clinical Trial Non Probability Convenient Sampling Technique Duration of treatment: 25 weeks 2 groups; (group A=30) SSAET +Normal routine medication+ Normal Dietary Plan , Other group (Group B=30) with normal routine medication + Normal Dietary Plan.

Patients will be enrolled in experimental group according to speeds test.

HYPOTHESIS:

Alternate hypothesis:

There is difference on the effects of Supervised Structured Aerobic Exercise Training Program on serum BDNF, androgens level, menstrual irregularity and quality of life in females with insulin resistant polycystic ovarian syndrome.

Null Hypothesis:

There is no difference on the effects of Supervised Structured Aerobic Exercise Training Program on serum BDNF, androgens level, menstrual irregularity and quality of life in females with insulin resistant polycystic ovarian syndrome.

OBJECTIVES:

To determine the effects of Supervised Structured Aerobic Exercise Training Program on quality of life in women with PCOS.

2. To determine the effect of Supervised Structured Aerobic Exercise Training Program on BDNF levels in women with PCOS.

3. To determine the effect of Supervised Structured Aerobic Exercise Training Program on mental health (stress, depression, anxiety) in women with PCOS.

4. To determine the effect of Supervised Structured Aerobic Exercise Training Program on BMI in women with PCOS.

5. To determine the effect of Supervised Structured Aerobic Exercise Training Program on menstrual irregularity in women with PCOS.

6. To determine the effect of Supervised Structured Aerobic Exercise Training Program on Aerobic fitness in women with PCOS.

7. To determine the effect of Supervised Structured Aerobic Exercise Training Program on androgens level in PCOS.

8. To determine the effect of Supervised Structured Aerobic Exercise Training Program on Lipid accumulation product in PCOS.

9. To determine the effect of Supervised Structured Aerobic Exercise Training Program on Glycemic control in PCOS.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome is a very common systemic disease consisting of hormone problem for women of childbearing age. Women with PCOS may not ovulate, have high levels of androgens, and have many small cysts on the ovaries. PCOS can cause missed or irregular menstrual periods, excess hair growth, acne, infertility, and weight gain. BDNF is linked with exercise and its receptors are also in ovaries. Hence, if the levels of BDNF falls below average then it plays an important role in hyperandrogenism and this often accompanied with lack of physical activity. Another factor, lipid accumulation product is closely related to glucose intolerance and wight gain which eventually gives rise to hyperandrogenism and it eventually affects the quality of life of females with polycystic ovarian syndrome.

It will be a randomized controlled trial. Convenient sampling technique would be used.

Inclusion criteria would be females of age 18-35 years, insulin resistant polycystic ovarian syndrome, pre-diagnosed, married and un married both, diabetic & nulliparous females.

Exclusion criteria would be post pill, Inflammatory & Adrenal PCOS, any psychological disease or disorder, any systemic disease other than PCOS (cushing syndrome, thyroid dysfunction, renal tumor, etc), Orthopedic conditions (including fracture, dislocation, etc), any surgery in past 6 months, involved in any other exercise regimen at the same time, having any specialized diet plan & Pregnant females.

Patients enrolled in the study will be divided randomly by even odd method. (Group A=30) will be given the Supervised Structured Aerobic Exercise Treatment Program for 12 weeks along with their normal routine medications given to them by their gynecologist.

(Group B=30) will have the conventional treatment of only the routine medications given by their gynecologist and brisk walk plan. Assessment of variables would be taken from both groups at baseline, 12 weeks and 25 weeks of intervention. 2 ml of blood would be taken through syringe and plasma would be tested for BDNF levels through ELISA, Androgens level through Free Androgen Index and quality of Life through Polycystic Ovarian Syndrome Quality of Life Questionnaire (PCOSQ). Aerobic fitness through Canadian fitness test and VO2max. Glycated hemoglobin would be tested for glucose intolerance through HbA1c test.

Keywords: Polycystic ovary syndrome, Poly cystic ovarian syndrome, sclerocystic ovaries, aerobic fitness, aerobic exercise, supervised, hyperandrogenism, PCOS, SHBG, testosterone, Quality of life.

HYPOTHESIS:

Alternate hypothesis:

There is difference on the effects of Supervised Structured Aerobic Exercise Training Program on serum BDNF, androgens level, menstrual irregularity and quality of life in females with insulin resistant polycystic ovarian syndrome.

Null Hypothesis:

There is no difference on the effects of Supervised Structured Aerobic Exercise Training Program on serum BDNF, androgens level, menstrual irregularity and quality of life in females with insulin resistant polycystic ovarian syndrome.

STUDY GROUPS:

Group 1: (Experimental Group n=30) Conventional Drugs treatment of PCOS advised by the medical specialist along with the Supervised Structured Aerobic Exercise Training program (SSAET) for 25 weeks.(29) Speed of the treadmill will be calculated and maintained at 60 to 70% of MHR in each session with progression of duration and inclination only. The intervention in experimental group would be divided into 5 phases of 5 weeks duration each.

DURATION OF EXERCISE SESSION

The patients in experimental group would be treated for a single session per day, at 3 days per week for 25 weeks. The details of each phase are given below:

Phase-1: In first phase the duration of each session would be 10 minutes and the total duration of exercise will be 30 minutes per week.

Phase-2: In the second phase the duration of a single session would be 20 minutes and duration21 of exercise per week will be 60 minutes.

Phase-3: In the third phase the duration of a single session would be 30 minutes and the total duration of exercise per week will be 90 minutes.

Phase-4: In the fourth phase the duration of each phase would be 40 minutes and the total duration of exercise per week will be 120 minutes.

Phase-5: In the last phase and final phase the duration of a single session would be 50 minutes and the total duration of exercise will be 150 minutes per week, as recommended by the American heart Association (AHA).

INCLINATION OF TREADMILL WALKING RAMP WITH GROUND (30) Phase-1: Normal Phase-2: 3 degrees Phase-3: 6 degrees Phase-4: 9 degrees Phase-5: 12 degrees Intensity of progression would be measured by the subject's Borgs rate of perceived exertion (RPE) according to the 15-point Borg Scale as per individual load.

Warm up and cool down protocol:

1. Without treadmill: warm up protocol involves breathing exercises, Stretching exercises (pectoralis major, triceps, biceps, hamstrings & calf stretch) and cool down exercises as ankle-toe movements of 5-10 min duration.
2. On tread mill: the warming-up phase, which consisted in walking on the treadmill for 5 minutes at low intensity (30% of MHR), at a 0% slope before the actual phase, and the cooling phase, which consist of in walking on the treadmill for 5 minutes at low intensity (30% of MHR) at 0% slope in each session. The MHR would be calculated according to the equation (HR= 220-age).

Group 2: (Control Group n=30) Conventional Drugs treatment of PCOS advised by the medical specialist along with the simple sustained brisk walk advised at a self-selected brisk pace described as "faster than normal walking but a pace that could be sustained for at least 20 min." Subjects would be instructed to complete at least three walks per week, each walk of 20 to 60 min duration.

TOOLS:

1. Modified polycystic ovarian syndrome Quality of Life Questionnaire (MPCOSQ)- Quality of life
2. MIQ (Menstrual Irregularity Questionnaire)- Menstrual irregularity
3. Women's weight in kilograms divided by the square of height in meters- BMI
4. Aerobic fitness- I. Canadian home fitness test, bench test from 8cm for 3 min II. Indirect estimation of VO2 max by formula VO2 max (walking) = (0.2 x speed of treadmill) + (0.9 x speed x treadmill grade) + 3.5
5. BDNF levels- ELISA
6. Androgens level- Serum SHBG will be measured by coated-tube immunoradiometric assay using commercial kits. Testosterone will be measured by RIA using commercial enzymatic kits. Free androgen index (FAI) will be calculated as testosterone/SHBG × 100.

   Clinical hyperandrogenism (a score of 6 or higher on the modified Ferriman-Gallwey scale)
7. Mental health- (Stress, depression & Anxiety) by DASS
8. Lipid Accumulation Product -Triglycerides test and waist circumference The LAP would be calculated as [waist circumference (centimeters) - 58] × [triglycerides (millimoles per liter)]
9. Glycemic control-HbA1c levels (Pre-diabetic condition as HbA1c 5.7-6.4% according to American Diabetic Association)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 To 35 years Females.
* Insulin resistant PCOS type.
* Already Diagnosed patients form gynecological department according to the Rotterdam criteria.
* Both Married and unmarried females.
* Nulliparous females.

Exclusion Criteria:

* Post pill PCOS, Inflammatory PCOS & Adrenal PCOS
* Any psychological disease or disorder
* Any systemic disease other than PCOS (cushing syndrome, thyroid dysfunction, etc)
* Orthopedic conditions (including fracture, dislocation, etc)
* Any surgery in past 6 months.
* Involved in any other exercise regimen at the same time.
* Having any specialized diet plan.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females only who are diagnosed by the gynecologist with polycystic ovarian syndrome according to Rotterdum criteria of diagnosing PCOS.
Enrollment: 60 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale (DASS) | 12 weeks and 25 weeks
  Mental Health (Stress, depression & Anxiety) by DASS 21
  Scoring Process:
  1. Sum the scores for each subscale:
     Add the scores for the 7 items within each subscale (Depression, Anxiety, and Stress).
  2. Multiply by 2:
     Multiply the sum of each subscale by 2 to get the final score for each area (Depression, Anxiety, and Stress).
  3. Interpret the scores:
  The resulting scores are then interpreted using the provided severity levels for each subscale.
  Severity Levels:
  The DASS-21 provides severity levels for each subscale:
  Depression:
  Normal (0-9), Mild (10-13), Moderate (14-20), Severe (21-27), Extremely Severe (28+).
  Anxiety:
  Normal (0-7), Mild (8-9), Moderate (10-14), Severe (15-19), Extremely Severe (20+).
  Stress:
  Normal (0-14), Mild (15-18), Moderate (19-25), Severe (26-33), Extremely Severe (34+).
  > Higher the scores means more severity and less healthy.
Polycystic ovarian syndrome Quality of Life Questionnaire (PCOSQOL) | 12 weeks and 25 weeks
  This is a tool to measure quality of life in females with Polycystic Ovarian syndrome.
  There are total 35 Questions in it. Scoring: Summate each item to give a total score. A low score represents that a lower quality of life, a higher score represents a lesser to no impact on quality of life.
MIQ (Menstrual Irregularity Questionnaire) | 12 weeks and 25 weeks
  Measures menstrual irregularity The MIQ is a 6-point questionnaire, and the total score reflects the overall impact of heavy menstrual bleeding on the woman's life. Higher scores indicate a greater negative impact of heavy menstrual bleeding on the woman's quality of life. The MIQ helps healthcare professionals understand the severity of the problem and tailor treatment accordingly.
3 min bench step test II. Indirect estimation of VO2 max by formula VO2 max (walking) = (0.2 x speed of treadmill) + (0.9 x speed x treadmill grade) + 3.5 | 12 weeks and 25 weeks
  To measure Aerobic fitness.
  YMCA 3-minute Bench Step Test:
  You step up and down on a 30 cm (12-inch) step for three minutes at a consistent pace, and your heart rate is measured afterward to estimate fitness for 1 minute through carotid artery. The more fit you are, the lower your recovery heart rate will be, meaning a lower number is a better score.
  Compare to Charts:
  Use your age and gender to find the appropriate fitness rating chart, such as the YMCA charts.
  Determine Your Level:
  The chart will show whether your 1-minute heart rate falls into categories like excellent, good, above average, average, or below average fitness.
  YMCA FEMALES Scoring:
  Excellent <109 Above Average 110 - 117 Average 118 - 134 Below Average 135-137 Poor >137
ELISA | 12 and 25 weeks
  BDNF levels
Androgens level | 12 weeks and 25 weeks
  Serum SHBG will be measured by coated-tube immunoradiometric assay using commercial kits. Testosterone will be measured by RIA using commercial enzymatic kits. Free androgen index (FAI) will be calculated as testosterone/SHBG × 100.
  Clinical hyperandrogenism (a score of 6 or higher on the modified Ferriman-Gallwey scale)

SECONDARY OUTCOMES:
HOMA-IR for Glycemic control | 12 weeks and 25 weeks
  The HOMA-IR score is calculated using your fasting glucose and fasting insulin levels:
  HOMA-IR = (Fasting Glucose x Fasting Insulin) / 22.5
Lipid Accumulation Product | 12 weeks and 25 weeks
  Triglycerides test and waist circumference The LAP would be calculated as [waist circumference (centimeters) - 58] × [triglycerides (millimoles per liter)]
BMI | 12 weeks and 25 weeks
  Women's weight in kilograms divided by the square of height in meters

CONTACTS AND LOCATIONS:
Overall Officials: Muzna Munir, ppdpt, Principal Investigator — Riphah International University
Locations (1):
- Sculpture Gym, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shakil-Ur-Rehman S, Karimi H, Gillani SA. Effects of supervised structured aerobic exercise training program on fasting blood glucose level, plasma insulin level, glycemic control, and insulin resistance in type 2 diabetes mellitus. Pak J Med Sci. 2017 May-Jun;33(3):576-580. doi: 10.12669/pjms.333.12023. PMID 28811774
- See also: Intervention being used on the other metabolic disorder — https://pubmed.ncbi.nlm.nih.gov/28811774/
- See also: Aerobic general exercises were applied for 12 weeks only to see the results on inflammatory markers. — https://pubmed.ncbi.nlm.nih.gov/35647831/
- See also: Relation of abnormal BDNF levels and PCOS — https://pubmed.ncbi.nlm.nih.gov/22420627/
- Available data/document: Study Protocol: PMID: 28811774 — https://pubmed.ncbi.nlm.nih.gov/28811774/ — Intervention is being used on other metabolic disorder. And the main principal investigator is the co-supervisor of the current research and i have taken the permission.

DOCUMENTS (4):
  • Study Protocol: ethical letter (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT07157371/Prot_000.pdf
  • Study Protocol and Statistical Analysis Plan: all detailed protocol. (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT07157371/Prot_SAP_001.pdf
  • Statistical Analysis Plan: statistical anaylsis (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT07157371/SAP_002.pdf
  • Informed Consent Form (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT07157371/ICF_003.pdf